CLINICAL TRIAL: NCT00546351
Title: A Multi-center, Open-label, follow-on Trial to Assess the Long-term Safety and Efficacy of Lacosamide in Subjects With Painful Distal Diabetic Neuropathy Including a Double-blind, Randomized Time Point Withdrawal Subtrial.
Brief Title: Study Evaluating Long-term Safety and Efficacy of Lacosamide in Subjects With Painful Distal Diabetic Neuropathy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0746; 2004-000551-42 (EudraCT Number)
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Results first posted 2012-04-19 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Painful Diabetic Neuropathy
Keywords: Lacosamide
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): 50 to 100 mg Lacosamide film-coated tablets; two times per day up to 600 mg/day; 6.5 years.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — 50 to 100 mg Lacosamide film-coated tablets; two times per day up to 600 mg/day; 6.5 years
  Other Names: Vimpat

SUMMARY:
SP746 (NCT00546351) is a multi-center, open-label, follow-on trial. The purpose of this trial is to assess safety and tolerability of long-term exposure of lacosamide (previously referred to as SPM 927) in subjects with painful distal diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed Study SP743 (NCT00238524) or SP874 (NCT00350103) and, in the investigator's opinion, might benefit from long-term administration of SP746 (NCT00546351). Exception: subjects who prematurely discontinued
* SP743 (NCT00238524) or SP874 (NCT00350103) due to lack of efficacy or due to intolerability to trial medication (after Visit 5but prior to entering the Maintenance Phase) may be eligible to participate in SP746 (NCT00546351), after consultation with the medical monitor

Exclusion Criteria:

* Subject has clinically relevant ECG abnormalities, or a QTc interval ≥500 ms, and/or a QTc interval increase of ≥60 ms from the mean pre-dose QTc value at Visit 2 of SP743 (NCT00238524) or SP874 (NCT00350103)
* Subject has aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≥3 times the upper limit of the normal range (ULN) with total bilirubin ≥2 times ULN or transaminases (AST and/or ALT) ≥5 times ULN
* Subject has a clinically relevant medical condition that, in the opinion of the investigator, jeopardizes or compromises the subject's ability to participate in this trial
* Subject is a pregnant or nursing female, or is of childbearing potential and is not surgically sterile, 2 years postmenopausal, or does not practice 2 combined methods of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2004-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (101):
- Austria (2):
  - 180, Vienna
  - 183, Vienna
- Belgium (6):
  - 003, Antwerp
  - 006, Bonheiden
  - 002, Genk
  - 001, Leuven
  - 005, Merksem
  - 004, Roeselare
- Bulgaria (10):
  - 011, Pleven
  - 014, Plovdiv
  - 017, Plovdiv
  - 019, Rousse
  - 012, Sofia
  - 013, Sofia
  - 015, Sofia
  - 016, Sofia
  - 210, Stara Zagora
  - 010, Varna
- Czechia (8):
  - 028, Brno
  - 220, Chomutov
  - 026, Litoměřice
  - 027, Olomouc
  - 024, Ostrava-Poruba
  - 029, Písek
  - 021, Prague
  - 022, Prague
- 192, Kuopio, Finland
- France (2):
  - 034, Lisieux
  - 031, Nevers
- Germany (22):
  - 040, Bad Saarow
  - 052, Beckum
  - 049, Berlin
  - 051, Berlin
  - 056, Berlin
  - 242, Berlin
  - 249, Berlin
  - 247, Bochum
  - 041, Hamburg
  - 045, Hamburg
  - 054, Hamburg
  - 244, Jena
  - 058, Köthen
  - 043, Künzing
  - 050, Leipzig
  - 053, Leipzig
  - 250, Leipzig
  - 046, Mittweida
  - 243, München
  - 246, Schwerin
  - 044, Stuhr-Brinkum
  - 248, Witten
- Hungary (11):
  - 060, Budapest
  - 062, Budapest
  - 061, Győr
  - 262, Kecskemét
  - 260, Makó
  - 266, Nyíregyháza
  - 064, Szeged
  - 265, Székesfehérvár
  - 264, Szolnok
  - 263, Tatabánya
  - 261, Veszprém
- Italy (3):
  - 270, Pavia
  - 273, Pavia
  - 272, Pozzilli
- Poland (14):
  - 092, Bialystok
  - 293, Bialystok
  - 094, Bydgoszcz
  - 095, Częstochowa
  - 091, Gdansk
  - 093, Gdansk
  - 294, Krakow
  - 297, Krakow
  - 090, Lodz
  - 295, Lodz
  - 291, Radom
  - 292, Warsaw
  - 296, Warsaw
  - 290, Ząbkowicki
- Romania (7):
  - 100, Bucharest
  - 102, Bucharest
  - 107, Bucharest
  - 108, Bucharest
  - 109, Bucharest
  - 101, Cluj-Napoca
  - 103, Timișoara
- Russia (5):
  - 114, Moscow
  - 115, Moscow
  - 116, Moscow
  - 112, Saint Petersburg
  - 111, Samara
- Serbia (4):
  - 140, Belgrade
  - 143, Belgrade
  - 144, Belgrade
  - 142, Niš
- 137, Granada, Spain
- United Kingdom (5):
  - 159, Bath
  - 154, Bristol
  - 152, Leeds
  - 150, Morriston
  - 151, Newport

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in May 2004 with subjects from Austria, Belgium, Bulgaria, Czech Republic, Finland, France, Germany, Hungary, Italy, Poland, Romania, Russia, Serbia, Spain, and United Kingdom. The primary completion date occurred in January 2011, with study completion in January 2011.
Pre-assignment Details: Participant Flow and Baseline Characteristics refer to the Safety Set (SS).
Period: Overall Study
Arm/Group | Lacosamide
Started | 621
Completed | 385
Not Completed | 236
Not completed — Adverse Event | 76
Not completed — Lack of Efficacy | 15
Not completed — Withdrawal by Subject | 109
Not completed — Lost to Follow-up | 9
Not completed — Protocol Deviation | 1
Not completed — Unsatisfactory compliance | 9
Not completed — Other reasons for premature termination | 17

BASELINE CHARACTERISTICS:
Arm/Group | Lacosamide
Number analyzed (Participants) | 621
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 500
  >=65 years | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 296
  Male | 325
Region of Enrollment [Number; unit: participants]
  Serbia | 54
  Finland | 1
  Spain | 2
  Austria | 9
  Russian Federation | 30
  United Kingdom | 19
  Italy | 7
  France | 6
  Czech Republic | 57
  Hungary | 76
  Belgium | 19
  Poland | 101
  Romania | 61
  Bulgaria | 62
  Germany | 117

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing the Occurrence of at Least One Treatment-emergent Adverse Event (TEAE) During the Evaluation Period From Entry Visit 1 Through End of Treatment (Approximately 6.5 Years).
Description: Adverse events are any untoward medical occurrences in a subject administered study treatment, whether or not these events are related to treatment.
Time Frame: From entry Visit 1 through end of treatment (approximately 6.5 years)
Population: This analysis includes all subjects (all 621) in the Safety Set (SS).
Measure: Number; unit: participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 621
participants | 416

2. Primary Outcome: Number of Participants Experiencing the Occurrence of at Least One Serious Adverse Event (SAE) During the Evaluation Period From Entry Visit 1 Through End of Treatment (Approximately 6.5 Years).
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Is fatal
  * Is life-threatening
  * Results in persistent or significant disability/incapacity
  * Requires inpatient hospitalization
  * Prolongs existing inpatient hospitalization
  * Is a congenital anomaly/birth defect
  * Is considered to be an important medical event. Such an event may not be immediately life threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the definitions above
Time Frame: From entry Visit 1 through end of treatment (approximately 6.5 years)
Population: This analysis includes all subjects (all 621) in the Safety Set (SS).
Measure: Number; unit: participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 621
participants | 132

3. Secondary Outcome: Average Daily Pain Score Using an 11-point Likert Scale (0-10) at Baseline Visit.
Description: On the Likert Scale, 0 = no pain and 10 = worst possible pain.
Time Frame: Baseline
Population: Of the 621 subjects in the Safety Set (SS), 620 are included in this analysis.
  Data was not available for 1 subject at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 620
units on a scale | 6.45 (1.371)

4. Secondary Outcome: Average Daily Pain Score Using an 11-point Likert Scale (0-10) at Last Visit.
Description: On the Likert Scale, 0 = no pain and 10 = worst possible pain.
Time Frame: Last Visit (approximately 2 years)
Population: Of the 621 subjects in the Safety Set (SS), 619 are included in this analysis.
  Data was not available for 2 subjects at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 619
units on a scale | 3.01 (2.246)

5. Secondary Outcome: Average Pain Score as Measured by a 100 mm Visual Analog Scale (VAS) at Baseline.
Description: Visual Analog Scale (VAS) 0 mm = no pain and 100 mm = worst possible pain.
Time Frame: Baseline
Population: Of the 621 subjects in the Safety Set (SS), 213 are included in this analysis.
  Data was not available for 408 subjects at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 213
units on a scale | 65.83 (15.986)

6. Secondary Outcome: Average Pain Score as Measured by a 100 mm Visual Analogue Scale (VAS) at Last Visit.
Description: On VAS 0 mm = no pain and 100 mm = worst possible pain.
Time Frame: Last Visit (approximately 2 years)
Population: Of the 621 subjects in the Safety Set (SS), 214 are included in this analysis.
  Data was not available for 407 subjects at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 214
units on a scale | 30.47 (23.940)

7. Secondary Outcome: Patient's Global Impression of Change (PGIC) at Last Visit.
Description: The PGIC is a 7-point self-administered categorical rating scale in which the subject rated the change in pain since starting trial medication (from much worse [score of 1] to much better [score of 7]).
  Reported results are presented as Better (sum of mildly, moderately, or much better), No Change, or Worse (sum of mildly, moderately, or much worse).
Time Frame: Last Visit (approximately 2 years)
Population: Of the 621 subjects in the Safety Set (SS), 551 are included in this analysis.
  Data was not available for 70 subjects at the time of this measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide
Number analyzed (Participants) | 551
percentage of participants
  Better | 82.6
  No Change | 11.4
  Worse | 6.0

8. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Intensity at Last Visit.
Description: 0 = no pain and 10 = most intense pain sensation imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: Of the 621 subjects of the Safety Set (SS), 195 are included in this analysis.
  Data was not available for 426 subjects at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 195
units on a scale | -3.2 (2.38)

9. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Sharpness at Last Visit.
Description: 0 = not sharp and 10 = most sharp sensation imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: Of the 621 subjects in the Safety Set (SS), 195 are included in this analysis.
  Data was not available for 426 subjects at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 195
units on a scale | 3.0 (2.23)

10. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Heat at Last Visit.
Description: 0 = not hot and 10 = the most hot sensation imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 195
units on a scale | 2.9 (2.35)

11. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Cold at Last Visit.
Description: 0 = not cold and 10 = the coldest sensation imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 195
units on a scale | 2.1 (2.19)

12. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Dullness at Last Visit.
Description: 0 = not dull and 10 = most dull sensation imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 195
units on a scale | 2.9 (2.11)

13. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Unpleasantness at Final Visit.
Description: 0 = not unpleasant and 10 = most unpleasant sensation imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: Of the 621 subjects in the Safety Set (SS), 193 are included in this analysis.
  Data was not available for 428 subjects at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 193
units on a scale | 3.8 (2.24)

14. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Surface Pain at Last Visit.
Description: 0 = no surface pain and 10 = most intense surface pain imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 193
units on a scale | 3.2 (2.17)

15. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Deep Pain at Last Visit.
Description: 0 = no deep pain and 10 = most intense deep pain imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 193
units on a scale | 3.4 (2.39)

16. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Itchiness at Final Visit.
Description: 0 = not itchy and 10 = most itchy sensation imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 195
units on a scale | 2.0 (2.06)

17. Secondary Outcome: Within-Subject Change in Neuropathic Pain Using the Neuropathic Pain Scale (NPS) - Sensitivity at Last Visit.
Description: 0 = not sensitive and 10 = most sensitive sensation imaginable.
Time Frame: Baseline Visit; Last Visit (approximately 2 years)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 195
units on a scale | 2.9 (2.31)

18. Secondary Outcome: Average Pain Interference With Sleep (11-point Likert Scale) at Baseline.
Description: 0 = no interference with sleep and 10 = worst possible interference with sleep.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 620
units on a scale | 5.98 (1.850)

19. Secondary Outcome: Average Pain Interference With Sleep (11-point Likert Scale) at Last Visit.
Description: 0 = no interference with sleep and 10 = worst possible interference with sleep.
Time Frame: Last Visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 619
units on a scale | 2.73 (2.281)

20. Secondary Outcome: Average Pain Interference With Activity (11-point Likert Scale) at Baseline.
Description: 0 = no interference with activity and 10 = worst possible interference with activity.
Time Frame: Baseline
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 620
units on a scale | 6.11 (1.660)

21. Secondary Outcome: Average Pain Interference With Activity (11-point Likert Scale) at Last Visit.
Description: 0 = no interference with activity and 10 = worst possible interference with activity.
Time Frame: Last Visit
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 619
units on a scale | 2.89 (2.349)

22. Secondary Outcome: Average Quality of Life Using the SF-36 Health Survey - Physical Component Summary (PCS) at Baseline.
Description: The SF-36 Health Survey measures health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores: PCS = physical functioning, role-physical, bodily pain, and general health; MCS = vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0 = worst score (or quality of life) and 100 = best score.
Time Frame: Baseline
Population: Of the 621 subjects in the Safety Set (SS), 588 are included in this analysis.
  Data was not available for 33 subjects at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 588
units on a scale | 32.8 (8.04)

23. Secondary Outcome: Average Quality of Life Using the SF-36 Health Survey - Physical Component Summary (PCS) at Last Visit.
Description: as for outcome 22
Time Frame: Last Visit
Population: Of the 621 subjects in the Safety Set (SS), 552 are included in this analysis.
  Data was not available for 69 subjects at the time of this measurement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 552
units on a scale | 38.4 (9.41)

24. Secondary Outcome: Average Quality of Life Using the SF-36 Health Survey - Mental Component Summary (MCS) at Baseline.
Description: as for outcome 22
Time Frame: Baseline
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 588
units on a scale | 42.8 (11.04)

25. Secondary Outcome: Average Quality of Life Using the SF-36 Health Survey - Mental Component Summary (MCS) at Last Visit.
Description: as for outcome 22
Time Frame: Last Visit
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lacosamide
Number analyzed (Participants) | 552
units on a scale | 44.5 (10.90)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from Entry Visit 1 through End of Treatment (Approximately 6.5 Years).
Description: Adverse Events refer to the Safety Set (SS). SS includes all subjects that were administered the investigational products at least once.
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 132/621
Other Adverse Events (participants affected / at risk) | 169/621
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=621)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 6 (6)
Coronary artery disease (Cardiac disorders) | 5 (5)
Myocardial infarction (Cardiac disorders) | 3 (3)
Bundle branch block right (Cardiac disorders) | 2 (2)
Bundle branch block left (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 2 (4)
Hypertensive cardiomyopathy (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Spondylolisthesis (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 5 (5)
Retinal haemorrhage (Eye disorders) | 1 (2)
Retinal detachment (Eye disorders) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (2)
Eye haemorrhage (Eye disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Perforated ulcer (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 2 (2)
Gangrene (Infections and infestations) | 2 (2)
Superinfection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Bronchitis fungal (Infections and infestations) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (2)
Erysipelas (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
QRS axis abnormal (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (8)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (12)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (6)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Toe deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Epithelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Loss of consciousness (Nervous system disorders) | 2 (3)
Presyncope (Nervous system disorders) | 2 (2)
Diabetic neuropathy (Nervous system disorders) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Drop attacks (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Apallic syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Brain stem syndrome (Nervous system disorders) | 1 (1)
Psychosomatic disease (Psychiatric disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Knee operation (Surgical and medical procedures) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)
Intermittent claudication (Vascular disorders) | 2 (2)
Circulatory collapse (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 2 (2)
Venous thrombosis limb (Vascular disorders) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 1 (1)
Diabetic macroangiopathy (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Arterial stenosis limb (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=621)
Vertigo (Ear and labyrinth disorders) | 34 (44)
Nasopharyngitis (Infections and infestations) | 49 (63)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (41)
Dizziness (Nervous system disorders) | 45 (49)
Headache (Nervous system disorders) | 38 (45)
Hypertension (Vascular disorders) | 40 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.